CLINICAL TRIAL: NCT01342133
Title: Sweat Duct Imaging in Mother/Newborn Dyads
Status: Completed | Type: Observational
Sponsor: Edimer Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ECP-005
Record Dates: First submitted 2011-04-22; First posted 2011-04-27 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: X-Linked Hypohidrotic Ectodermal Dysplasia
MeSH Terms: conditions — Ectodermal Dysplasia 1, Anhidrotic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Newborns
- Mothers

SUMMARY:
The purpose of this study is to evaluate sweat duct number on the plantar surface of newborn infants using a non-invasive confocal microscopy device.

DETAILED DESCRIPTION:
In this exploratory study, the investigators propose to evaluate sweat duct number on the plantar surface of newborn infants using a non-invasive confocal microscopy device (Lucid Vivascope®). This approach has the potential to be valuable in repeated sweat endpoint assessments, as the device was selected based on its ease of use, the low risk to patients of all ages, and its ability to generate quantitative data.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term newborns (37-42 weeks gestation at delivery) in the Assessment Nursery at Barnes-Jewish Hospital, St. Louis, MO
* Mother of a healthy term newborn who is enrolled in this study

Exclusion Criteria:

* Congenital abnormalities affecting skin, nails, or hair in the newborn infant
* Family history of a sweating disorder

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll up to twenty healthy term newborns and their mothers in the Assessment Nursery at Barnes-Jewish Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2011-04; Primary Completion 2011-04 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Demonstrate the use of a confocal microscope to quantify sweat ducts on the plantar surface of healthy, term newborns | Day 1
  To demonstrate the ease of use of a non-invasive confocal imaging device in the evaluation and measurement of sweat ducts on the plantar surface of healthy, term newborns. These measurements will be used as comparison data in subsequent trials involving those affected by X-Linked Hypohidrotic Ectodermal Dysplasia.
To assess the sweat duct density (i.e. the number of sweat ducts) in a 6 x 6 mm area on the plantar surface of healthy, term newborns, males and females, and the palmar surface of their mothers | Day 1
  These measurements will be used as comparison data in subsequent trials involving those affected by X-Linked Hypohidrotic Ectodermal Dysplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Moscoso, MD, PhD, Principal Investigator — Washington University School of Medicine; Dorothy K Grange, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States